CLINICAL TRIAL: NCT04779060
Title: Intrathecal Fentanyle Versus Dexamethasone in Patients Under Going Gynacological Laparoscopic Surgeries
Brief Title: Intrathecal Fentanyle Versus Dexamethasone in Gynacological Laparoscopic Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, lecturer of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13700331
Record Dates: First submitted 2021-02-27; First posted 2021-03-03 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Intraoperativ Pain
MeSH Terms: interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fentanyle group (Active Comparator)
  Interventions: Drug: intrathecal fentanyle
- dexamethasone group (Active Comparator)
  Interventions: Drug: dexamethasone
- control group (Placebo Comparator)
  Interventions: Drug: saline

INTERVENTIONS:
Drug: intrathecal fentanyle — 25 mic fentanyle added to heavy bupivacaine for spinal anesthesia
  Arms: fentanyle group
Drug: dexamethasone — 8 mg dexamethasone give intrathecally for spinal anaesthesia
  Arms: dexamethasone group
Drug: saline — normal saline will be mixed with bupivacaine intrathecally
  Arms: control group

SUMMARY:
Laparoscopy was first introduced to the medical field of in the middle of the last century. It revolutionized the surgical interventions; it reduced the total medical expenditures and hastened postoperative recovery . General anaesthesia (GA) was considered the only anesthetic technique suitable for laparoscopic interventions, and several myths and facts prevented regional anaesthesia (RA) implementation. Respiratory and Cardiovascular impairment were the main aspects of concern which are thought to be best controlled by GA

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II
* elective gynacological laparoscopic surgery

Exclusion Criteria:

* patient refusal
* chronic kidney and hepatic diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
intraoperative pain | 60 minutes
  pain measured by VAS score =from 0 to 10 0-3 is mild pain 3-6 moderate pain 6-10 sever pain

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt